CLINICAL TRIAL: NCT03586973
Title: A Phase 2, Open-Label, Single-Arm Study of Cabozantinib in Japanese Patients With Advanced Hepatocellular Carcinoma Who Have Received Prior Systemic Anticancer Therapy
Brief Title: A Phase 2 Study of Cabozantinib in Japanese Participants With Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cabozantinib-2003; U1111-1214-6141 (Other: WHO); JapicCTI-184018 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2018-06-29; First posted 2018-07-16 (Actual); Results first posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Advanced Hepatocellular Carcinoma
MeSH Terms: interventions — cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A: Cabozantinib 60 mg (Experimental): Participants who have received first/second line anticancer therapy with sorafenib were assigned to Cohort A and received cabozantinib 60 milligrams (mg), tablet, orally, once daily in the fasted state, up to approximately 2 years.
  Interventions: Drug: Cabozantinib
- Cohort B: Cabozantinib 60 mg (Experimental): Participants who did not receive first/second line anticancer therapy with sorafenib were assigned to Cohort B and received cabozantinib 60 mg, tablet orally, once daily in the fasted state, up to approximately 2 years.
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — Cabozantinib tablet
  Other Names: XL184

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of cabozantinib in Japanese participants with advanced hepatocellular carcinoma (HCC) who have received prior systemic anticancer therapy.

DETAILED DESCRIPTION:
The drug being tested in this study is called Cabozantinib. Cabozantinib is being tested to treat advanced hepatocellular carcinoma in Japanese patients. This study will look at the efficacy and safety of Cabozantinib.

The study will enroll approximately 34 patients. Participants will be assigned to Cohort A (at least 17 participants) or Cohort B (approximately 15 participants) and will receive the following treatment. Participants who have received prior sorafenib will enroll to Cohort A and participants who have not received prior sorafenib will enroll to Cohort B.

- Cabozantinib 60 mg

All participants will be asked to take one tablet of cabozantinib once daily in the fasted state (dose at least 2 hours after meal and no more food intake for 1 hour postdose) throughout the study.

This multi-center trial will be conducted in Japan. The overall time to participate in this study is approximately at most 3 years. Participants will make multiple visits to the clinic during the treatment and posttreatment period, including a follow-up assessment after last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female Japanese participants 20 years of age or older on the day of consent.
2. Histological or cytological diagnosis of HCC (results of a previous biopsy will be accepted).
3. Measurable disease per response evaluation criteria in solid tumors (RECIST) 1.1 as determined by the investigator.
4. Participants who have disease that is not amenable to a curative treatment approach (eg, transplant, surgery, radiofrequency ablation).
5. Participants who have received 1 or 2 prior anticancer therapies for advanced HCC.

   * Cohort A: participants who have received prior sorafenib.
   * Cohort B: participants who have not received prior sorafenib. Note: Additional prior systemic therapies used as adjuvant or local therapy are allowed.
6. Radiographic progression following prior systemic anticancer therapy for advanced HCC.
7. Recovery to =<Grade 1 Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03 from toxicities related to any prior treatments, unless the Adverse Events (AEs) are clinically nonsignificant and/or stable on supportive therapy.
8. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1, and life expectancy of at least 3 months.
9. Child-Pugh Score of A.
10. Adequate organ and marrow function at Screening (within 10 days before Week 1 Day 1):

    1. Absolute neutrophil count (ANC) >=1,200/mm^3.
    2. Platelets >=60,000/mm^3.
    3. Hemoglobin >=8 g/dL.
    4. Serum creatinine =<1.5 × upper limit of normal (ULN) or calculated creatinine clearance >=40 mL/min using the Cockroft-Gault equation.
    5. Urine protein-to-creatinine ratio (UPCR) =<1 mg/mg Cr.
    6. Total bilirubin =<2 mg/dL.
    7. Serum albumin >=2.8 g/dL.
    8. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =<5.0 × ULN.
    9. Hemoglobin A1c (HbA1c) =<8% (if HbA1c results are unavailable [eg, hemoglobin variant], a fasting serum glucose =<160 mg/dL).
11. Antiviral therapy per local standard of care if active hepatitis B virus (HBV) infection.
12. Female participants who:

    1. Are postmenopausal (natural amenorrhea, not due to other medical reasons) for at least 1 year before the Screening visit, OR
    2. Are surgically sterile, OR
    3. If they are of childbearing potential, agree to practice 1 highly effective method of birth control with a condom, which is an effective barrier method of contraception, at the same time, from the time of signing the informed consent through 4 months after the last dose of study drug, OR
    4. Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant, from the time of signing the informed consent through 4 months after the last dose of study drug. (Periodic abstinence [eg, calendar, ovulation, symptothermal, postovulation methods], condoms only, withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception.)

       Male participants, even if surgically sterilized (ie, status postvasectomy), who:
    5. Agree to practice effective barrier contraception during the entire study treatment period and through 4 months after the last dose of study drug. If their partner are of childbearing potential, their female partner should use 1 highly effective method of birth control at the same time, OR
    6. Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant, from the time of signing the informed consent through 4 months after the last dose of study drug. (Periodic abstinence [eg, calendar, ovulation, symptothermal, postovulation methods for the female partner], condoms only, withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception.)
13. Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the participant at any time without prejudice to future medical care.
14. Participant is willing and able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

1. Fibrolamellar carcinoma or mixed hepatocellular cholangiocarcinoma.
2. Any type of anticancer agent within 14 days before the first day of study drug administration (Week 1 Day 1).
3. Radiation therapy within 28 days (14 days for radiation for bone metastases) or radionuclide treatment (eg, I-131 or Y-90) within 42 days before Week 1 Day 1 (participant is excluded if there are any clinically relevant ongoing complications from prior radiation therapy).
4. Prior Cabozantinib treatment.
5. Treatment with any investigational products (excluding anticancer products approved in Japan) within 28 days before Week 1 Day 1.
6. Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 3 months before Week 1 Day 1. Eligible participants must be without corticosteroid treatment at Week 1 Day 1.
7. Concomitant anticoagulation, with oral anticoagulants (eg, warfarin, direct thrombin and Factor Xa inhibitors) or platelet inhibitors (eg, clopidogrel).

   Note: Low-dose aspirin for prophylactic use (per local applicable guidelines) and low-dose, low molecular weight heparins (LMWH) are permitted (LMWH has not been approved for the use for cardioprotection in Japan). Anticoagulation with therapeutic doses of LMWH is allowed in participants without radiographic evidence of brain metastasis, who are on a stable dose of LMWH for at least 12 weeks before Week 1 Day 1, and who have had no complications from a thromboembolic event or the anticoagulation regimen.
8. Participants who have uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

   1. Cardiovascular disorders including

      * Symptomatic congestive heart failure, unstable angina pectoris, or serious cardiac arrhythmias.
      * Uncontrolled hypertension defined as sustained blood pressure (BP) >150 mm Hg systolic, or >100 mm Hg diastolic despite optimal antihypertensive treatment.
      * Stroke (including transient ischemic attack [TIA]), myocardial infarction, or other ischemic event within 6 months before Week 1 Day 1.
      * Thromboembolic event within 3 months before Week 1 Day 1.
      * A left-ventricular ejection fraction =<50%.
   2. Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation:

      * Tumors invading the GI tract, active peptic ulcer disease, inflammatory bowel disease (eg, Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis or acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction.
      * Abdominal fistula, GI perforation, bowel obstruction, intra-abdominal abscess within 6 months before Week 1 Day 1.

      Note: Complete healing of an intra-abdominal abscess must be confirmed prior to Week 1 Day 1.
   3. Major surgery within 2 months before Week 1 Day 1. Complete healing from major surgery must have occurred 1 month before Week 1 Day 1. Complete healing from minor surgery (eg, simple excision, tooth extraction) must have occurred at least 7 days before Week 1 Day 1. Participants with clinically relevant complications from prior surgery are not eligible.
   4. Cavitating pulmonary lesion(s) or endobronchial disease.
   5. Lesion invading a major blood vessel including, but not limited to: inferior vena cava, pulmonary artery, or aorta. Participants with invasion or thromboses of portal/hepatic vasculature attributed to underlying liver disease and/or liver tumor are eligible.
   6. Clinically significant bleeding risk including the following within 3 months before Week 1 Day 1: hematuria, hematemesis, hemoptysis of >0.5 teaspoon (>2.5 mL) of red blood, or other signs indicative of pulmonary hemorrhage, or history of other significant bleeding if not due to reversible external factors.
   7. Other clinically significant disorders such as:

      * Active infection requiring systemic treatment.
      * Known infection with human immunodeficiency virus, or known acquired immunodeficiency syndrome -related illness.
      * Active hepatitis B and/or C. Participants with active hepatitis virus infection controlled with antiviral therapy are eligible.
      * Serious non-healing wound/ulcer/bone fracture.
      * Malabsorption syndrome.
      * Uncompensated/symptomatic hypothyroidism.
      * Requirement for hemodialysis or peritoneal dialysis.
      * History of solid organ transplantation.
9. Participants with untreated or incompletely treated varices with bleeding or high risk for bleeding. Participants treated with adequate endoscopic therapy (according to institutional standards) without any episodes of recurrent GI bleeding requiring transfusion or hospitalization for at least 6 months before Week 1 Day 1 are eligible.
10. Moderate or severe ascites.
11. Corrected QT interval calculated by the Fridericia formula (QTcF) >500 msec within 14 days before Week 1 Day 1.

    Note: If the QTcF is >500 msec in first electrocardiogram (ECG), a total of 3 ECGs each separated by at least 3 minutes should be performed within 30 minutes. If the average of these 3 consecutive results for QTcF is =<500 msec, the participant meets eligibility in this regard.
12. Inability to swallow tablets.
13. Previously identified allergy or hypersensitivity to components of the study treatment formulations.
14. Female participants who are lactating and breastfeeding or have a positive serum pregnancy test during the Screening period.

    Note: Female participants who are in the lactation period, even if they discontinue breastfeeding, will be excluded from the study.
15. Previously diagnosed with another malignancy and have any evidence of residual disease within 2 years before Week 1 Day 1.

    Note: Participants with superficial skin cancers, or localized, low-grade tumors deemed cured and not treated with systemic therapy are not excluded.
16. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
17. Known GI disease or GI procedure that could interfere with the oral absorption or tolerance of Cabozantinib.
18. Use of strong cytochrome P450 (CYP) 3A inhibitors and CYP3A inducers within 14 days before Week 1 Day 1.
19. Admission or evidence of illicit drug use, drug abuse, or alcohol abuse.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2021-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (17):
- Japan (17):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Iizuka Hospital, Iizuka, Fukuoka
  - Kurume University Hospital, Kurume, Fukuoka
  - Sapporo-Kosei General Hospital, Sapporo, Hokkaido
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Kindai University Hospital, Sayama, Osaka
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Kyorin University Hospital, Mitaka, Tokyo
  - Japanese Red Cross Musashino Hospital, Musashino, Tokyo
  - Chiba University Hospital, Chiba
  - Hiroshima University Hospital, Hiroshima
  - Okayama University Hospital, Okayama
  - Osaka City University Hospital, Osaka
  - Osaka International Cancer Institute, Osaka

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Kudo M, Tsuchiya K, Kato N, Hagihara A, Numata K, Aikata H, Inaba Y, Kondo S, Motomura K, Furuse J, Ikeda M, Morimoto M, Achira M, Kuroda S, Kimura A. Cabozantinib in Japanese patients with advanced hepatocellular carcinoma: a phase 2 multicenter study. J Gastroenterol. 2021 Feb;56(2):181-190. doi: 10.1007/s00535-020-01753-0. Epub 2021 Jan 3. PMID 33392749

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 15 investigative sites in Japan from 06 August 2018 to 29 June 2021.
Pre-assignment Details: Participants with a diagnosis of advanced hepatocellular carcinoma (HCC) were enrolled in this study in two Cohorts A and B. Participants who received prior sorafenib were enrolled in Cohort A and participants who received prior systemic anticancer therapy other than sorafenib were enrolled in Cohort B.
Period: Overall Study
Arm/Group | Cohort A: Cabozantinib 60 mg | Cohort B: Cabozantinib 60 mg
Started | 20 | 14
Completed | 0 | 0
Not Completed | 20 | 14
Not completed — Death | 15 | 8
Not completed — Site Terminated by Sponsor | 3 | 6
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Cabozantinib 60 mg | Cohort B: Cabozantinib 60 mg | Total
Number analyzed (Participants) | 20 | 14 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.2 (6.32) | 71.6 (8.13) | 72 (7.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 17 | 14 | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 20 | 14 | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 20 | 14 | 34
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 20 | 14 | 34
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 162.2 (8.31) | 165.4 (7.08) | 163.5 (7.88)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 61.60 (9.123) | 64.54 (11.351) | 62.81 (10.042)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] — Body Mass Index=weight (kg)/[height (m)^2]
  kilogram per square meter (kg/m^2) | 23.34 (2.262) | 23.46 (2.894) | 23.39 (2.5)
History of Drinking Alcohol [Count of Participants; unit: Participants] — Participants were divided as per the history of drinking alcohol.
  Participants
    Current Drinker | 6 | 5 | 11
    Former Drinker | 10 | 9 | 19
    Never Drunk | 4 | 0 | 4
Current Etiology of Disease [Count of Participants; unit: Participants] — Participants were divided as per the etiology of disease at baseline. Participants were counted more than once in multiple categories. The current etiology (cause of disease or condition) is reported in categories as: 1) Hepatitis B (Without Hepatitis C), 2) Hepatitis C (Without Hepatitis B), 3) Hepatitis B and C, 4) Hepatitis B (Regardless of Hepatitis C), 5) Hepatitis C (Regardless of Hepatitis B), 6) Without Hepatitis B and C, 7) Alcoholism, 8) Nonalcoholic Steatohepatitis (NASH), 8) Other
  Participants
    Hepatitis B (Without Hepatitis C) | 5 | 1 | 6
    Hepatitis C (Without Hepatitis B) | 7 | 3 | 10
    Hepatitis B and C | 0 | 1 | 1
    Hepatitis B (Regardless of Hepatitis C) | 5 | 2 | 7
    Hepatitis C (Regardless of Hepatitis B) | 7 | 4 | 11
    Without Hepatitis B and C | 8 | 9 | 17
    Alcoholism | 5 | 5 | 10
    Nonalcoholic Steatohepatitis (NASH) | 1 | 2 | 3
    Other | 3 | 2 | 5
Child-Pugh Score: Grade A [Count of Participants; unit: Participants] — Child-Pugh score was graded as A to C based on total score from Points assigned, where A- well-compensated disease; B- significant functional compromise; C-decompensated disease. Data is reported for those categories with at least one participant.
  Participants | 20 | 14 | 34
Extrahepatic Spread and/or Macrovascular Invasion [Count of Participants; unit: Participants]
  Presence | 7 | 6 | 13
  No presence | 13 | 8 | 21
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS): Grade 1 [Count of Participants; unit: Participants] — The ECOG scale was as follows: Grade 0: Fully active, able to perform all pre-disease activities without restriction; Grade 1: Restricted in physically strenuous activity, ambulatory, able to carry out light work; Grade 2: Ambulatory and capable of all self-care but unable to work. Up and about more than 50% of waking hours; Grade 3: Capable of only limited self-care, confined to bed or chair > 50% of waking hours; Grade 4: Completely disabled. Cannot carry on any self-care. Only categories with participants are reported.
  Participants | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: 24-Week Progression-Free Survival Rate (PFSR)
Description: 24-week PFSR=percentage of participants with progression-free survival (PFS) of at least 24 weeks at Week 25 Day 1 plus 7 days. PFS=time from first day of study drug administration to earlier of progressive disease (PD) or death due to any cause per Response Evaluation Criteria in Solid Tumors Version 1.1(RECIST 1.1). PD=at least a 20% increase in sum of target lesion diameters (SoD) with reference to smallest(nadir) SoD. In addition to relative increase of 20%, SoD must also demonstrate an absolute increase of at least 5 mm. For nontarget lesion time Point Response, unequivocal progression of nontarget lesions. Modest 'increase' in size of one or more nontarget lesions is usually not sufficient to quality for unequivocal progression status, it must not be representative of single lesion increase. Lesion in an anatomical location and not scanned at baseline is considered new lesion. Lesion qualifies as PD if finding is unequivocally not due to change in imaging technique or modality.
Time Frame: Week 25 Day 1 plus 7 days
Population: Full Analysis Set (FAS) included participants who received at least one dose of study drug.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: Cabozantinib 60 mg | Cohort B: Cabozantinib 60 mg
Number analyzed (Participants) | 20 | 14
percentage of participants | 59.8 [36.06 to 77.21] | 16.7 [4.02 to 36.82]

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as time from the first day of study drug administration to the earlier of PD per RECIST 1.1 as assessed by IRC or death due to any cause. Per RECIST 1.1, for target lesion time point response, PD was defined at least a 20% increase in the SoD of target lesions, taking as a reference the smallest (nadir) SoD since (and including) baseline. In addition to the relative increase of 20%, the SoD must also demonstrate an absolute increase of at least 5 mm. For nontarget lesion time point response, unequivocal progression of nontarget lesions. A modest 'increase' in the size of one or more nontarget lesions is usually not sufficient to quality for unequivocal progression status. It must be representative of overall disease status change, not a single lesion increase. The lesion qualifies as a PD if the finding is unequivocally not due to a change in the imaging technique or modality.
Time Frame: Until disease progression, or death or end of study (Up to approximately 2.8 years)
Population: FAS included participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A: Cabozantinib 60 mg | Cohort B: Cabozantinib 60 mg
Number analyzed (Participants) | 20 | 14
months | 7.4 [5.5 to 9.5] | 3.6 [1.8 to 5.6]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants whose best overall response was complete response (CR) or partial response (PR) per RECIST 1.1 as assessed by IRC, which was confirmed by a subsequent evaluation conducted >= 28 days later. Per RECIST 1.1, for target lesion time point response, CR was defined disappearance of all target lesions. All pathological lymph nodes (whether target or nontarget) must have reduction in short axis to <10 mm. For nontarget lesion time point response, disappearance of all nontarget lesions. All lymph nodes must be nonpathological in size (<10 mm short axis); PR was defined as at least a 30% decrease in SoD of target lesions, taking as a reference the baseline SoD.
Time Frame: Up to approximately 2 years
Population: FAS included participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: Cabozantinib 60 mg | Cohort B: Cabozantinib 60 mg
Number analyzed (Participants) | 20 | 14
percentage of participants | 5.0 [0.127 to 24.873] | 0.0 [0.000 to 23.164]

4. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR=percentage of participants whose best overall response is CR,PR or SD, per RECIST 1.1, CR and PR require confirmation by subsequent evaluation conducted >=28 days later, and SD have to be maintained for at least 8 weeks after first day of study drug administration. CR=disappearance of all target lesions. All pathological lymph nodes (whether target or nontarget) must have reduction in short axis to <10 mm. For nontarget lesion time point response, disappearance of all nontarget lesions. All lymph nodes must be nonpathological in size (<10 mm short axis); PR=at least a 30% decrease in SoD of target lesions, taking as reference baseline SoD; SD=neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD; SoD must also demonstrate an absolute increase of at least 5 mm; PD=at least a 20% increase in SoD of target lesions, taking as a reference smallest (nadir) SoD.
Time Frame: Up to approximately 2 years
Population: FAS included participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: Cabozantinib 60 mg | Cohort B: Cabozantinib 60 mg
Number analyzed (Participants) | 20 | 14
percentage of participants | 85.0 [62.107 to 96.793] | 64.3 [35.138 to 87.240]

5. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as time from the first day of study drug administration to death due to any cause. Participants without documentation of death were censored on the date they were last known to be alive.
Time Frame: Up to end of study (Up to approximately 2.8 years)
Population: FAS included participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A: Cabozantinib 60 mg | Cohort B: Cabozantinib 60 mg
Number analyzed (Participants) | 20 | 14
months | 19.3 [13.3 to 22.6] | 9.9 [3.6 to NA] — Upper limit of 95% confidence interval was not estimable due to lower number of participants with the event.

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: Up to end of study (Up to approximately 2.8 years); Serious and other adverse events: From first dose up to 30 days post last dose (Up to approximately 2 years)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Cohort A: Cabozantinib 60 mg | Cohort B: Cabozantinib 60 mg
All-Cause Mortality (participants affected / at risk) | 15/20 | 8/14
Serious Adverse Events (participants affected / at risk) | 7/20 | 2/14
Other Adverse Events (participants affected / at risk) | 20/20 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Cabozantinib 60 mg (N=20) | Cohort B: Cabozantinib 60 mg (N=14)
Gastrointestinal ulcer (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 1
Biloma (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Liver abscess (Infections and infestations) | 1 | 0
Meningitis bacterial (Infections and infestations) | 1 | 0
Peritonitis bacterial (Infections and infestations) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Cabozantinib 60 mg (N=20) | Cohort B: Cabozantinib 60 mg (N=14)
Anaemia (Blood and lymphatic system disorders) | 3 | 2
Lymphopenia (Blood and lymphatic system disorders) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 7 | 3
Dry eye (Eye disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 15 | 6
Constipation (Gastrointestinal disorders) | 1 | 6
Stomatitis (Gastrointestinal disorders) | 4 | 2
Vomiting (Gastrointestinal disorders) | 5 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 3 | 1
Ascites (Gastrointestinal disorders) | 2 | 1
Periodontal disease (Gastrointestinal disorders) | 1 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Anal erosion (Gastrointestinal disorders) | 0 | 1
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1
Glossodynia (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 5 | 3
Malaise (General disorders) | 6 | 2
Pyrexia (General disorders) | 3 | 4
Oedema peripheral (General disorders) | 3 | 1
Oedema (General disorders) | 2 | 0
Chest pain (General disorders) | 1 | 0
Influenza like illness (General disorders) | 0 | 1
Mass (General disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 3 | 2
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1
Seasonal allergy (Immune system disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 5 | 1
Bronchitis (Infections and infestations) | 0 | 1
Cystitis bacterial (Infections and infestations) | 1 | 0
Folliculitis (Infections and infestations) | 0 | 1
Fungal oesophagitis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 1 | 0
Periodontitis (Infections and infestations) | 1 | 0
Purulence (Infections and infestations) | 0 | 1
Tinea cruris (Infections and infestations) | 1 | 0
Tinea faciei (Infections and infestations) | 0 | 1
Tinea infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urethritis (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 2 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Skin injury (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Platelet count decreased (Investigations) | 6 | 7
Aspartate aminotransferase increased (Investigations) | 6 | 6
Alanine aminotransferase increased (Investigations) | 5 | 5
Neutrophil count decreased (Investigations) | 5 | 2
Blood thyroid stimulating hormone increased (Investigations) | 3 | 3
Weight decreased (Investigations) | 5 | 1
Blood lactate dehydrogenase increased (Investigations) | 3 | 2
Amylase increased (Investigations) | 3 | 1
Lipase increased (Investigations) | 1 | 2
White blood cell count decreased (Investigations) | 1 | 2
Blood alkaline phosphatase increased (Investigations) | 2 | 0
Blood creatinine increased (Investigations) | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Blood urine present (Investigations) | 0 | 1
Glomerular filtration rate decreased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0
Liver function test increased (Investigations) | 1 | 0
Neutrophil count increased (Investigations) | 1 | 0
Urine protein/creatinine ratio increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 8 | 7
Hyperammonaemia (Metabolism and nutrition disorders) | 3 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dysgeusia (Nervous system disorders) | 4 | 3
Headache (Nervous system disorders) | 2 | 0
Taste disorder (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 0
Proteinuria (Renal and urinary disorders) | 3 | 4
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Haemoglobinuria (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0
Breast mass (Reproductive system and breast disorders) | 1 | 0
Gynaecomastia (Reproductive system and breast disorders) | 1 | 0
Scrotal oedema (Reproductive system and breast disorders) | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 8 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 16 | 10
Rash (Skin and subcutaneous tissue disorders) | 3 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 9 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2018-10-30): https://cdn.clinicaltrials.gov/large-docs/73/NCT03586973/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-05): https://cdn.clinicaltrials.gov/large-docs/73/NCT03586973/SAP_001.pdf